CLINICAL TRIAL: NCT02687620
Title: Does Immunogenicity Have an Influence on the Efficacy of Anti-tumor Necrosis Factor (Anti-TNF) Therapy in Patients With Ankylosing Spondylitis (AS): An Inception Cohort Study
Brief Title: Does Immunogenicity Have an Influence on the Efficacy of Anti-TNF Therapy in Patients With AS: An Inception Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Dr. Servet Akar, Prof, Izmir Katip Celebi University
Other Study IDs: KCU-12032014
Record Dates: First submitted 2016-02-03; First posted 2016-02-22 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Ankylosing Spondylitis; Axial Spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the serum sample aquisition whole blood samples with EDTA will be collected and stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AS patients receiving Anti-TNF treatment: Three hundred and fifty consecutive AS patients fulfilling the modified New York criteria for the classification of AS (5), and with a new anti-TNF agent prescription (either for the first time or switched) in the last two weeks period will be included. Treatment with anti-TNF agents will be in accordance with the regulations of Turkish Social Security Agency (SGK) on the initiation and continuation of anti-TNF agents in AS, as well as ASAS/EULAR recommendations for the management of AS (29, 30).

SUMMARY:
The purpose of this prospective cohort study is to evaluate the influence of serum drug levels and development of anti-drug antibodies on clinical response to anti-TNF agents in ankylosing spondylitis(AS) treatment. Secondary aims are to assess the demographic, clinical and laboratory variables associated with the development of anti-TNF drug antibodies at baseline or disease course and to reveal the impact of anti-drug antibodies on long-term efficacy or safety in particular drug survival in AS patients treated in daily clinical practice.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic inflammatory rheumatic disease that predominantly affects sacroiliac joints and spine. It is the prototype of spondyloarthritides (SpA) and one of the most common rheumatic diseases. Sacroiliitis is the earliest manifestation of disease and accompanying with spinal involvement cause inflammatory back pain (IBP). IBP usually starts insidiously in the early adulthood and typically it is felt deep in the buttock and/or lower lumbar regions. It improves with activity and returns with the rest and is usually accompanied by morning stiffness lasting at least 30 minutes. Involvement of the spine in patients with AS is usually not limited to the sacroiliac joints and lumbar region and usually it extends up to the thoracic and cervical segment. Currently the only sign that is diagnostic for AS is radiographic sacroiliitis. However radiography detects structural changes and take up to ten years to appear unequivocally.

In some patients bone tenderness due to enthesitis may be the primary complaint. Arthritis in the hips and shoulders occur in some patients and is associated with worse prognosis. Typical arthritis pattern in AS patients is asymmetric and usually involves the lower extremity joints. There are several extra-articular features of AS and the most common is acute anterior uveitis.

Until recently treatment options for AS were limited and based on non-steroidal anti-inflammatory drugs (NSAIDs), traditional disease modifying anti-rheumatic drugs (DMARDs) for the rheumatoid arthritis and physical therapy. The last decade witnessed a major advance in AS therapy with the use of anti-tumor necrosis factor (anti-TNF) agents. Anti-TNF agents have a substantial effect not only the axial disease but also in peripheral arthritis, enthesitis and extra-articular features (like psoriasis and inflammatory bowel disease). Currently there are four anti-TNF agents approved for AS: (1) infliximab which is a monoclonal chimeric antibody and given at a dose of 5 mg/kg every 6-8 weeks; (2) etanercept which is human TNF receptor fusion protein and administered subcutaneously at a dose of 50 mg/once a week; (3) adalimumab which is a humanized monoclonal antibody and administered as subcutaneous injection at a dose of 40 mg fortnightly; and (4) golimumab which is a fully human monoclonal antibody and administered subcutaneously at a dose of 50 mg once a month.

Since there is no head-to-head studies comparing the anti-TNF agents in the treatment of AS patients there is no ranking for the prescription of anti-TNF agents. Mixed treatment comparisons (that is statistical model allowing the simultaneous multiple meta-analysis of different pair-wise comparisons) between infliximab, adalimumab and etanercept did not show a statistically significant difference. Indeed similar improvements in Bath ankylosing spondylitis activity index (BASDAI 50) scores and ASAS partial remission (between 45.2% to 51.0% BASDAI 50 and 22.1% to 22.4% for partial remission) have been reported in randomized controlled clinical trials.

Although many AS patients respond very well to anti-TNF therapy, a considerable amount of them do not and additionally a significant proportion of patients have to stop their treatment. In clinical practice the reported 1-year and 2-year drug survival rates for anti-TNF agents are 70-85% and 60-75%, respectively.Moreover in a substantial proportion of patients either increase in the administered dosage or dosing frequency have become necessary. Therefore factors, which can predict the response or related with the primary or secondary non-response for anti-TNF treatment have a growing attention among treating specialists. In a study providing an overview of clinical trials and observational studies showed that increased acute phase reactants, higher disease activity, functional status, younger age, and HLA-B27 positivity were independent baseline predictors of response to anti-TNF treatment and increased acute phase reactants, presence of peripheral arthritis, and male sex were the predictors of long-term drug survival.

Immunogenicity refers to development of antibodies by the adaptive immune system in response to foreign substances. The development of anti-drug antibodies were extensively studied in rheumatoid arthritis and it was shown that anti-drug antibodies has a varying impact on the clinical efficacy depending on whether these antibodies are neutralizing or non-neutralizing. Recent review demonstrated that neutralizing antibodies are associated with a reduced chance of achieving a minimal disease activity or clinical remission, decreased drug survival, increased dose escalation and adverse drug reactions in RA patients. However data regarding the immunogenicity in patients treated with AS is scarce and somewhat controversial. In a small study including 38 AS patients treated with infliximab de Vries et al showed that anti-infliximab antibodies was found significantly more often (59% vs 5%) and mean serum through infliximab levels were significantly lower in ASAS20 non-responders. In the above-mentioned study infusion reactions were also seemed to be associated with the development of anti-drug antibodies. In another study de Vries et al (26) were found no antibodies to etanercept and similar serum etanercept levels in responder and non-responder AS patients (n=53). Same group also observed that anti-adalimumab antibodies were become detectable in 31% of AS (n=35) patients in 6 months period and this corresponded with diminished serum drug levels.

Arends et al reported that 0 to 30% of AS patients (n=60) developed anti-drug antibodies during one year of follow-up of anti-TNF treatment and patients with anti-IFN or anti-ADA antibodies had significantly lower drug serum levels.

The objective of this prospective cohort study is to evaluate the influence of serum drug levels and development of anti-drug antibodies on clinical response to anti-TNF agents. The assessment of demographic, clinical and laboratory variables associated with the development of anti-TNF drug antibodies at baseline or disease course will be also evaluated. Via this study, it might also be possible to reveal the impact of anti-drug antibodies on long-term efficacy or safety in particular drug survival in AS patients treated in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients whom are receiving their first anti-TNF treatment(not switch)
* Ankylosing spondylitis diagnosis according to modified New York Criteria
* Patients whom were older than 18 years old on anti-TNF initiation

Exclusion Criteria:

* Spondyloarthritis other than AS
* HIV positive or malignancy
* Being treated with another biological drug prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three hundred and fifty consecutive AS patients fulfilling the modified New York criteria for the classification of AS, and with a new anti-TNF agent prescription (either for the first time or switched) in the last two weeks period will be included. Treatment with anti-TNF agents will be in accordance with the regulations of Turkish Social Security Agency (SGK) on the initiation and continuation of anti-TNF agents in AS, as well as ASAS/EULAR recommendations for the management of AS.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-09; Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Serum drug levels | 0, 3, 6 12 and 24 months of the study
  It will be measured in mg/L or other measurement levels by using ELISA
Anti-drug antibody levels | 0, 3, 6 12 and 24 months of the study
  It will be measured in AU/mL or other measurement levels by using ELISA

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | every third months up to 104 weeks
  In order to evaluate function BASDAI will be evaluated in numeric rating scale (0-10)
Bath Ankylosing Spondylitis Functional Index (BASFI) | every third months up to 104 weeks
  In order to evaluate function BASFI will be evaluated in numeric rating scale (0-10)
Ankylosing Spondylitis Disease Activity Index (ASDAS) | every third months (if available) up to 104 weeks
  ASDAS-CRP (the preferred version) will be calculated by using the following formula:
  0.12 X Back pain + 0.06 X Duration of morning stiffness + 0.11 X Patient global + 0.07 X Peripheral pain / swelling + 0.58 X Ln (CRP + 1)

CONTACTS AND LOCATIONS:
Overall Officials: Servet Akar, Prof, Principal Investigator — İzmir Katip Celebi University School of Medicine
Locations (13):
- Turkey (Türkiye) (13):
  - Cukurova University School of Medicine, Adana
  - Ankara İbn-i Sina University School of Medicine, Ankara
  - Gülhane Askeri Tıp Akademisi School of Medicine, Ankara
  - Hacettepe University School of Medicine, Ankara
  - Adnan Menderes University School of Medicine, Aydin
  - Fırat University School of Medicine, Elâzığ
  - Osman Gazi University School of Medicine, Eskişehir
  - Goztepe Training and Research Hospital, Istanbul
  - Istanbul University Cerrahpasa School of Medicine, Istanbul
  - Istanbul University Istanbul School of Medicine, Istanbul
  - Ege University School of Medicine, Izmir
  - İzmir Katip Celebi University School of Medicine, Izmir
  - Kocaeli University School of Medicine, Kocaeli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braun J, Bollow M, Remlinger G, Eggens U, Rudwaleit M, Distler A, Sieper J. Prevalence of spondylarthropathies in HLA-B27 positive and negative blood donors. Arthritis Rheum. 1998 Jan;41(1):58-67. doi: 10.1002/1529-0131(199801)41:13.0.CO;2-G. PMID 9433870
- [Background] Onen F, Akar S, Birlik M, Sari I, Khan MA, Gurler O, Ergor A, Manisali M, Akkoc N. Prevalence of ankylosing spondylitis and related spondyloarthritides in an urban area of Izmir, Turkey. J Rheumatol. 2008 Feb;35(2):305-9. Epub 2007 Dec 15. PMID 18085733
- [Background] Sieper J, Braun J, Rudwaleit M, Boonen A, Zink A. Ankylosing spondylitis: an overview. Ann Rheum Dis. 2002 Dec;61 Suppl 3(Suppl 3):iii8-18. doi: 10.1136/ard.61.suppl_3.iii8. PMID 12381506
- [Background] Burgos-Vargas R, Braun J. Inflammatory back pain. Rheum Dis Clin North Am. 2012 Aug;38(3):487-99. doi: 10.1016/j.rdc.2012.08.014. Epub 2012 Sep 14. PMID 23083750
- [Background] van der Linden S, Valkenburg HA, Cats A. Evaluation of diagnostic criteria for ankylosing spondylitis. A proposal for modification of the New York criteria. Arthritis Rheum. 1984 Apr;27(4):361-8. doi: 10.1002/art.1780270401. PMID 6231933
- [Background] Feldtkeller E, Khan MA, van der Heijde D, van der Linden S, Braun J. Age at disease onset and diagnosis delay in HLA-B27 negative vs. positive patients with ankylosing spondylitis. Rheumatol Int. 2003 Mar;23(2):61-6. doi: 10.1007/s00296-002-0237-4. Epub 2002 Sep 3. PMID 12634937
- [Background] Mau W, Zeidler H, Mau R, Majewski A, Freyschmidt J, Stangel W, Deicher H. Clinical features and prognosis of patients with possible ankylosing spondylitis. Results of a 10-year followup. J Rheumatol. 1988 Jul;15(7):1109-14. PMID 3262757
- [Background] Rudwaleit M, Khan MA, Sieper J. The challenge of diagnosis and classification in early ankylosing spondylitis: do we need new criteria? Arthritis Rheum. 2005 Apr;52(4):1000-8. doi: 10.1002/art.20990. No abstract available. PMID 15818678
- [Background] Braun J, Deodhar A, Dijkmans B, Geusens P, Sieper J, Williamson P, Xu W, Visvanathan S, Baker D, Goldstein N, van der Heijde D; Ankylosing Spondylitis Study for the Evaluation of Recombinant Infliximab Therapy Study Group. Efficacy and safety of infliximab in patients with ankylosing spondylitis over a two-year period. Arthritis Rheum. 2008 Sep 15;59(9):1270-8. doi: 10.1002/art.24001. PMID 18759257
- [Background] van der Heijde D, Kivitz A, Schiff MH, Sieper J, Dijkmans BA, Braun J, Dougados M, Reveille JD, Wong RL, Kupper H, Davis JC Jr; ATLAS Study Group. Efficacy and safety of adalimumab in patients with ankylosing spondylitis: results of a multicenter, randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2006 Jul;54(7):2136-46. doi: 10.1002/art.21913. PMID 16802350
- [Background] Arends S, Brouwer E, van der Veer E, Groen H, Leijsma MK, Houtman PM, Th A Jansen TL, Kallenberg CG, Spoorenberg A. Baseline predictors of response and discontinuation of tumor necrosis factor-alpha blocking therapy in ankylosing spondylitis: a prospective longitudinal observational cohort study. Arthritis Res Ther. 2011 Jun 20;13(3):R94. doi: 10.1186/ar3369. PMID 21689401
- [Background] Glintborg B, Ostergaard M, Krogh NS, Dreyer L, Kristensen HL, Hetland ML. Predictors of treatment response and drug continuation in 842 patients with ankylosing spondylitis treated with anti-tumour necrosis factor: results from 8 years' surveillance in the Danish nationwide DANBIO registry. Ann Rheum Dis. 2010 Nov;69(11):2002-8. doi: 10.1136/ard.2009.124446. Epub 2010 May 28. PMID 20511613
- [Background] Kristensen LE, Karlsson JA, Englund M, Petersson IF, Saxne T, Geborek P. Presence of peripheral arthritis and male sex predicting continuation of anti-tumor necrosis factor therapy in ankylosing spondylitis: an observational prospective cohort study from the South Swedish Arthritis Treatment Group Register. Arthritis Care Res (Hoboken). 2010 Oct;62(10):1362-9. doi: 10.1002/acr.20258. PMID 20506310
- [Background] Kristensen LE, Geborek P, Saxne T. Dose escalation of infliximab therapy in arthritis patients is related to diagnosis and concomitant methotrexate treatment: observational results from the South Swedish Arthritis Treatment Group register. Rheumatology (Oxford). 2009 Mar;48(3):243-5. doi: 10.1093/rheumatology/ken467. Epub 2008 Dec 23. PMID 19106164
- [Background] Alawadhi A, Alawneh K, Alzahrani ZA. The effect of neutralizing antibodies on the sustainable efficacy of biologic therapies: what's in it for African and Middle Eastern rheumatologists. Clin Rheumatol. 2012 Sep;31(9):1281-7. doi: 10.1007/s10067-012-2040-2. Epub 2012 Aug 9. PMID 22875700
- [Background] de Vries MK, Wolbink GJ, Stapel SO, de Vrieze H, van Denderen JC, Dijkmans BA, Aarden LA, van der Horst-Bruinsma IE. Decreased clinical response to infliximab in ankylosing spondylitis is correlated with anti-infliximab formation. Ann Rheum Dis. 2007 Sep;66(9):1252-4. doi: 10.1136/ard.2007.072397. Epub 2007 May 1. PMID 17472991
- [Background] de Vries MK, van der Horst-Bruinsma IE, Nurmohamed MT, Aarden LA, Stapel SO, Peters MJ, van Denderen JC, Dijkmans BA, Wolbink GJ. Immunogenicity does not influence treatment with etanercept in patients with ankylosing spondylitis. Ann Rheum Dis. 2009 Apr;68(4):531-5. doi: 10.1136/ard.2008.089979. Epub 2008 Mar 28. PMID 18375542
- [Background] de Vries MK, Brouwer E, van der Horst-Bruinsma IE, Spoorenberg A, van Denderen JC, Jamnitski A, Nurmohamed MT, Dijkmans BA, Aarden LA, Wolbink GJ. Decreased clinical response to adalimumab in ankylosing spondylitis is associated with antibody formation. Ann Rheum Dis. 2009 Nov;68(11):1787-8. doi: 10.1136/ard.2009.109702. No abstract available. PMID 19822712
- [Background] Arends S, Lebbink HR, Spoorenberg A, Bungener LB, Roozendaal C, van der Veer E, Houtman PM, Griep EN, Limburg PC, Kallenberg CG, Wolbink GJ, Brouwer E. The formation of autoantibodies and antibodies to TNF-alpha blocking agents in relation to clinical response in patients with ankylosing spondylitis. Clin Exp Rheumatol. 2010 Sep-Oct;28(5):661-8. Epub 2010 Oct 22. PMID 20822711
- [Background] Horne R, Weinman J. Patients' beliefs about prescribed medicines and their role in adherence to treatment in chronic physical illness. J Psychosom Res. 1999 Dec;47(6):555-67. doi: 10.1016/s0022-3999(99)00057-4. PMID 10661603